CLINICAL TRIAL: NCT06418243
Title: Non-interventional Study on the Contribution of 3D Modelling in Surgical Management of Pediatric Retroperitoneal and Pelvic Tumors Compared to 2D Imaging
Brief Title: Contribution of 3D Modeling in Surgical Management of Pediatric Retroperitoneal and Pelvic Tumors
Acronym: 3D-PEDSURG
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Imagine Institute (Other); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230680; 2023-A02070-45 (Other: ID-RCB)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Tumor; Retroperitoneal Tumor
Keywords: Surgery; 3D-Imaging; MRI; CT Scan; Paediatric surgery; Tumor
MeSH Terms: conditions — Pelvic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children planned to get an MRI or CT scan: Children with a pelvic or retroperitoneal tumor requiring an MRI or CT scan for a possible surgical intervention

SUMMARY:
This study's purpose is the comparison of the automatically segmented 3D model to the reference manual segmentation, based on the Dice precision index. It is implemented by making parents' patients, surgeons and surgical helpers answer specific questions comparing 3D images to usual 2D images of the patient's tumor.

DETAILED DESCRIPTION:
The investigator will inform the child and his parents during the pre-surgical consultation, and will collect their non-opposition to be included in the study at the latest on the day of the MRI examination or CT scan. Patients requiring emergency imaging will not be included.

Pelvic tumors will benefit from MRI imaging and renal tumors from MRI and/or CT scan.

A CT scan will be carried out for retroperitoneal tumors other than renal tumors (mainly neuroblastomas).

All of the above examinations are carried out as part of the usual treatment, in the month preceding the surgery.

Pre-operatively After the imaging has been carried out, the 2D images will be presented to the patient and his family before surgery as it is done routinely. The 3D image will be showed afterwards. The family will have the opportunity to ask questions which the surgeon will answer as usually done.

The specific questionnaire will be completed by the patient and his family at the end of the consultation and given to the research team.

Once the patient is included and the examinations have been carried out, the operating surgeons and their assistants (help No. 1 and 2) will look at the 2D images, followed by the 3D images secondly a few days before surgery. They will complete the specific questionnaire and give it to the research team.

Once the patient is included and the imaging examinations have been carried out, surgeons external to the service will be contacted by the research team to organize a remote review session. The 2D images will be presented to them first, followed by the 3D images on the visualization software, via a remote communication system with screen sharing. They will complete the specific questionnaire independently and a copy of the questionnaires will then be sent to the research team by email and the originals sent by post.

Intraoperatively:

The 3D model of the patient will be displayed in the operating room, and/or integrated into the robot's display console (for robot-assisted surgeries) during the surgical procedure. At the end of the surgery, the operating surgeon and his assistants will complete (independently) a questionnaire on the consistency of the 2D and 3D images with the anatomy identified during the procedure and on the help or not provided by the 3D model.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Children between 3 months and less than 18 years old
* Children with a pelvic tumor requiring an MRI for a possible surgical intervention
* Children with a retroperitoneal tumor requiring a CT scan or MRI with a view to surgical intervention
* Children with no contraindication for a CT scan and/or 3T MRI
* Children whose parents do not object to their participation in the study

Other participants:

* Operating surgeon agreeing to participate in the study
* Caregiver agreeing to participate in the study
* External surgeon agreeing to participate in the study

Exclusion Criteria:

Children :

* Contraindication to MRI: metallic ocular foreign body, pacemaker, mechanical heart valve, old vascular clips on cerebral aneurysm
* Need for an MRI under general anaesthesia
* Contraindication for a CT scan with injection: renal failure, allergy to iodinated contrast products
* Patients having participated in a therapeutic clinical trial involving a new molecule within 30 days before inclusion
* Emergency situation

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a pelvic or retroperitoneal tumor requiring an MRI or CT scan for a possible surgical intervention coming at the hospital for a consultation as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Segmentation comparison | 1 month
  Comparison of the automatically segmented 3D model to the reference manual segmentation, based on the Dice precision index

SECONDARY OUTCOMES:
Distance comparison | 1 month
  Distance comparison between the reference segmentation and the one obtained by the algorithm using the Hausdorff spacing.
Anatomical structure recognition comparison | Day 0
  Recognition of anatomical structures comparison from 2D imaging and 3D imaging from score 1/score 3 of the pré-operative questionnaire for operating or external surgeons
Pre-operative planning contribution | Day 0
  Contribution of 3D modeling comparison to 2D imaging in pre-operative planning from score 2/score 4 of the pre-operative questionnaire for operating or external surgeons
Added value evaluation | Day 0
  Added value evaluation of 3D modelling compared to 2D imaging by using score 5 of the pre-operative questionnaire for operating or external surgeons
Surgeons' support evaluation in pre-operative routine | Day 0
  Surgeons' support evaluation for integrating 3D modelling into routine pre-operative planning from score 6 of the pre-operative questionnaire for operating or external surgeons
2D imaging evaluation contribution for families' understanding | Day 0
  Evaluation of the contribution of 3D modelling for families in understanding the information (pathology and surgery) delivered by the surgeon to parents pre-operatively from score 1 of the family questionnaire
3D modelling evaluation contribution for families' understanding | Day 0
  Evaluation of the contribution of 3D modelling for families in understanding the information (pathology and surgery) delivered by the surgeon to parents pre-operatively from score 2 of the family questionnaire
3D modelling added value evaluation pre-operatively | Day 0
  Added value evaluation of 3D modelling compared to 2D imaging for families pre-operatively from score 3 of the family questionnaire
3D modelling added value evaluation during surgery | 1 month
  Contribution of 3D modelling evaluation compared to 2D imaging for surgeons during surgery from score 1 of the post-operative questionnaire for operating surgeons and their helpers
Consistency evaluation between 3D modelling and anatomy | 1 month
  Consistency evaluation of the 3D imaging with anatomy observed intraoperatively from score 2 of the post-operative questionnaire for operating surgeons and their helpers
Surgeons' support evaluation in current practice | 1 month
  Surgeons' support evaluation for integrating 3D modeling into their current practice from score 3 of the post-operative questionnaire for operating surgeons and their helpers

CONTACTS AND LOCATIONS:
Overall Officials: Sabine SARNACKI, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wake N, Wysock JS, Bjurlin MA, Chandarana H, Huang WC. "Pin the Tumor on the Kidney:" An Evaluation of How Surgeons Translate CT and MRI Data to 3D Models. Urology. 2019 Sep;131:255-261. doi: 10.1016/j.urology.2019.06.016. Epub 2019 Jun 22. PMID 31233814
- [Background] Talanki VR, Peng Q, Shamir SB, Baete SH, Duong TQ, Wake N. Three-Dimensional Printed Anatomic Models Derived From Magnetic Resonance Imaging Data: Current State and Image Acquisition Recommendations for Appropriate Clinical Scenarios. J Magn Reson Imaging. 2022 Apr;55(4):1060-1081. doi: 10.1002/jmri.27744. Epub 2021 May 27. PMID 34046959
- [Background] Ibrahim I, Skoch A, Herynek V, Jiru F, Tintera J. Magnetic resonance tractography of the lumbosacral plexus: Step-by-step. Medicine (Baltimore). 2021 Feb 12;100(6):e24646. doi: 10.1097/MD.0000000000024646. PMID 33578590
- [Background] van der Zee JM, Fitski M, Simonis FFJ, van de Ven CP, Klijn AJ, Wijnen MHWA, van der Steeg AFW. Virtual Resection: A New Tool for Preparing for Nephron-Sparing Surgery in Wilms Tumor Patients. Curr Oncol. 2022 Feb 1;29(2):777-784. doi: 10.3390/curroncol29020066. PMID 35200565
- [Background] Bertrand MM, Macri F, Mazars R, Droupy S, Beregi JP, Prudhomme M. MRI-based 3D pelvic autonomous innervation: a first step towards image-guided pelvic surgery. Eur Radiol. 2014 Aug;24(8):1989-97. doi: 10.1007/s00330-014-3211-0. Epub 2014 May 17. PMID 24838739
- [Background] Simons DC, Buser MAD, Fitski M, van de Ven CP, Ten Haken B, Wijnen MHWA, Tan CO, van der Steeg AFW. Multi-modal 3-Dimensional Visualization of Pediatric Neuroblastoma: Aiding Surgical Planning Beyond Anatomical Information. J Pediatr Surg. 2024 Aug;59(8):1575-1581. doi: 10.1016/j.jpedsurg.2024.02.025. Epub 2024 Feb 24. PMID 38461108
- [Background] Valls-Esteve A, Adell-Gomez N, Pasten A, Barber I, Munuera J, Krauel L. Exploring the Potential of Three-Dimensional Imaging, Printing, and Modeling in Pediatric Surgical Oncology: A New Era of Precision Surgery. Children (Basel). 2023 May 3;10(5):832. doi: 10.3390/children10050832. PMID 37238380
- [Background] Hampshire J, Dicken BJ, Uruththirakodeeswaran T, Punithakumar K, Noga M. Pediatric patient-specific three-dimensional virtual models for surgical decision making in resection of hepatic and retroperitoneal tumors. Int J Comput Assist Radiol Surg. 2023 Oct;18(10):1941-1949. doi: 10.1007/s11548-023-02852-y. Epub 2023 Mar 11. PMID 36905500
- [Background] Bernhard JC, Isotani S, Matsugasumi T, Duddalwar V, Hung AJ, Suer E, Baco E, Satkunasivam R, Djaladat H, Metcalfe C, Hu B, Wong K, Park D, Nguyen M, Hwang D, Bazargani ST, de Castro Abreu AL, Aron M, Ukimura O, Gill IS. Personalized 3D printed model of kidney and tumor anatomy: a useful tool for patient education. World J Urol. 2016 Mar;34(3):337-45. doi: 10.1007/s00345-015-1632-2. Epub 2015 Jul 11. PMID 26162845
- [Background] Youn JK, Park SJ, Choi YH, Han JW, Ko D, Byun J, Yang HB, Kim HY. Application of 3D printing technology for pre-operative evaluation, education and informed consent in pediatric retroperitoneal tumors. Sci Rep. 2023 Jan 30;13(1):1671. doi: 10.1038/s41598-023-28423-4. PMID 36717595